CLINICAL TRIAL: NCT04047953
Title: The Study of Paclitaxel (Albumin-bound) Combined With Oxaliplatin and S-1 Conversion Therapy for Initial Unresectable Local Advanced or Potentially Resectable Metastatic Gastric Adenocarcinoma
Brief Title: Paclitaxel (Albumin-bound) Combined With Oxaliplatin and S-1 Conversion Therapy for Gastric Adenocarcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Zhaode Bu, Clinical Professor, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC-conversion
Record Dates: First submitted 2019-08-06; First posted 2019-08-07 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Gastric Adenocarcinoma
Keywords: Paclitaxel (albumin-bound); gastric cancer; conversion therapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Paclitaxel; Oxaliplatin; S 1 (combination); 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Conversion Therapy (Experimental): Paclitaxel (albumin-bound) +S-1+Oxaliplatin
  Interventions: Drug: Paclitaxel (albumin-bound) combined with Oxaliplatin and S-1

INTERVENTIONS:
Drug: Paclitaxel (albumin-bound) combined with Oxaliplatin and S-1 — Paclitaxel (albumin-bound) : 150 mg/m2, iv,d1. S-1 : 40~60mg，bid, d1-14( BSA<1.25m2，40mg；1.25m2≤BSA≤1.5m2，50mg；BSA>1.5m2，60mg) Oxaliplatin: 85mg/m2, iv, d1. Twenty-one days per cycle, a total of four cycles, after two cycles of treatment, the tumor was evaluated. The clinical efficacy was evaluated as CR\PR\SD and decided by the investigator to continue the treatment for two cycles or directly.
  Other Names: Paclitaxel (albumin-bound) + Oxaliplatin + S-1; Nab-paclitaxel + Oxaliplatin + S-1

SUMMARY:
To evaluate the efficacy and safety of Paclitaxel (albumin-bound) combined with Oxaliplatin and S-1 conversion therapy for initial unresectable local progression or potential resectable metastatic gastric adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18-75 years; male or female.
* Karnofsky Performance Status Score ≥70.
* Histological diagnosis of gastric adenocarcinoma, HER2 expression negative.
* The initial unresectable locally advanced or potentially resectable metastatic gastric adenocarcinoma, potentially resectable factor includes a single liver metastases, localized abdominal para-aortic lymph node (16a1 / b2) metastasis or positive abdominal free cancer cells.
* Physical condition and organ function allow for larger abdominal surgery.
* Subject baseline blood routine and blood biochemistry indexes meet the following criteria: hemoglobin(HB) ≥90 g/L; absolute neutrophil count(ANC) ≥1.5×109 /L; platelet count(PLT) ≥100×109 /L; alanine glutamate transaminase (ALT) and glutamate transaminase (AST) ≤2.5 x upper limit of normal range (ULN); total bilirubin (TBIL)≤1.5 x upper limit of normal range (ULN); Creatinine(Cr)≤1.5 x upper limit of normal range(ULN); Serum albumin≥30g/L.
* Echocardiographic scan confirmed left ventricular ejection fraction (LVEF) ≥ 50%.
* No serious accompanying disease lead to a survival period of <5 years.
* Agree and be able to follow the protocol during the study period.
* Written informed consent was provided prior to the study screening and the patient was informed that the study could be withdrawn at any time during the study without any loss.

Exclusion Criteria:

* For the treatment of the gastric cancer, patients who have received cytotoxic chemotherapy, radiotherapy or immunotherapy, except corticosteroids.
* Pregnancy or breastfeeding woman.
* Women of childbearing age who had a positive pregnancy test at baseline or who did not undergo a pregnancy test. Menopausal women must be stopped for at least 12 months to ensure that no pregnancy is possible.
* Men and women who have sex (with fertility probability) are reluctant to contraception during the study.
* Patients with ascites and positive abdominal free cancer cells.
* There are other history of malignant disease in the last 5 years, except for cured skin cancer and cervical carcinoma in situ.
* Those with a history of epilepsy, central nervous system disease, or mental disorder may be judged by the investigator that their clinical severity may hinder the signing of informed consent or affect the patient's oral medication compliance.
* Clinically severe (active) heart disease, such as symptomatic coronary heart disease, New York Heart Association (NYHA) class II or more severe congestive heart failure or severe drug-affected arrhythmias, or there is a history of myocardial infarction in the last 12 months.
* Upper gastrointestinal stagnation or abnormal physiological function or malabsorption syndrome may affect the absorption of S-1.
* It is known to have peripheral neuropathy ≥ NCI CTC AE grade 2. However, only the deep sputum reflex (DTR) disappears and the patient does not have to be excluded.
* Organ transplantation requires immunosuppressive therapy.
* Severe uncontrolled recurrent infections, or other serious uncontrolled concomitant diseases.
* Moderate or severe renal impairment [creatinine clearance equal to or lower than 50ml/min (calculated according to Cockcroft and Gault equations), or serum creatinine > upper normal limit (ULN).
* Those suffering from dihydropyrimidine dehydrogenase (DPD) deficiency are known.
* Those who are allergic to taxanes or any research ingredients.
* Those who received research medications or preparations/treatments (ie, participated in other trials) within 4 weeks prior to enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2019-09-10 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | within 4 weeks following the operation
  Proportion of patients who achieved R0 resection

SECONDARY OUTCOMES:
Progression free survival (PFS) | 5 years
  the time from registration to the date of disease progression or death resulting from any cause.
overall survival (OS) | 5 years
  the time from registration to the date of death resulting from any cause or the last follow-up visit.
Adverse Events(AEs) | until 28 days after the last study drug administration
  AEs are evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jiafu ji, MD, Principal Investigator — Peking University Cancer Hospital & Institute; Zhaode Bu, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China